CLINICAL TRIAL: NCT01219517
Title: Validation of the Accuracy of DNA Fingerprinting Using Polar Bodies and Embryonic Cells
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Reproductive Medicine Associates of New Jersey (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None
Other Study IDs: RMA-00-18
Record Dates: First submitted 2010-10-08; First posted 2010-10-13 (Estimated); Last update posted 2013-01-23 (Estimated); Status verified 2013-01

CONDITIONS: DNA Fingerprinting
Keywords: IVF; embryo biopsy; DNA fingerprinting; SNP

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Study Group (Experimental): All patients in the study receive the same treatment. All will have 2 polar body biopsies and all embryos biopsied prior to transfer.
  Interventions: Other: Polar body and embryo biopsy

INTERVENTIONS:
Other: Polar body and embryo biopsy — 2 polar bodies and all embryos will be biopsied prior to embryo transfer.
  Other Names: embryo biospy; SNP

SUMMARY:
The purpose of this study is to validate the ability to assess the genetic differences (DNA fingerprinting) on polar bodies (excess genetic material given off from the egg) and cells so that this technique may be used in the future to confirm markers of reproductive competence and improve the efficiency and safety of clinical human in vitro fertilization.

DETAILED DESCRIPTION:
Our group has recently validated a technique involving whole genomic amplification followed by single nucleotide polymorphisms (SNP) analysis which allows DNA fingerprinting of single cells. Given that there are more than 3.3 billion base pairs that constitute the human genome, there are approximately 3 million sites where routine variation in the genetic code exists. These SNPs have been identified on average to occur approximately once every 1000 base pairs (bp) and are present on all chromosomes.

100 couples will undergo routine in vitro fertilization (IVF) stimulation, the protocol to be determined by the patient's primary doctor. Following oocyte retrieval and intracytoplasmic sperm injection (ICSI), the first polar body will be biopsied using standard laboratory procedures, and sent for genetic analysis. 24 hours later, the second polar body will be biopsied and sent for genetic analysis. Finally, the embryos will be biopsied prior to transfer and the cell will be sent for gentic analysis. Genetic results are not available prior to transfer and there are be no delays in the treatment schedule as a result of the study. Buccal swabs are collected from infants. SNP profiles are created from the polar body and embryo biopsies which are then compared to the SNP profiles created from the buccal swabs.

ELIGIBILITY:
Major Inclusion: The following are major inclusion criteria:

1. Maximum of one prior failed IVF treatment cycle
2. Female partner less than 43 years of age
3. Normal day 3 FSH level (<12 mIU/mL)
4. Basal antral follicle count greater than or equal to 8
5. Ejaculated sperm specimen from the male partner with greater than 100,000 total motile
6. Donor sperm okay if patient is willing to purchase 3 extra vials for DNA testing

Exclusions: The following are exclusion criteria:

1. Diagnosis of chronic anovulation secondary to polycystic ovarian disease
2. Diagnosis of endometrial insufficiency
3. Clinical indication for PGD
4. Testicular biopsy or aspiration procedures to obtain sperm

Ages: 21 Years to 43 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 100 (Actual)
Dates: Start 2008-01; Primary Completion 2009-05 (Actual); Study Completion 2009-12 (Actual)

PRIMARY OUTCOMES:
Validate DNA fingerprinting | After delivery of infant(s)
  Comparison of the SNP profile from the buccal swab as compared to the SNP profile of the 1st polar body biopsy, the SNP profile of the 2nd polar body biopsy and the SNP profile of the embryo biopsy will show which biopsy provides the greatest predictive value of the DNA of the conceptus.

CONTACTS AND LOCATIONS:
Overall Officials: Richard T Scott, MD, Principal Investigator — Reproductive Medicine Associates of New Jersey
Locations (6):
- United States (6):
  - Colorado Center for Reproductive Medicine, Lone Tree, Colorado
  - Reproductive Medicine Associates of Connecticut, Norwalk, Connecticut
  - Reproductive Medicine Associates of Michigan, Troy, Michigan
  - Reproductive Medicine Associates, Morristown, New Jersey
  - Reproductive Medicine Associates of Vassar Brothers, Fishkill, New York
  - Reproductive Medicine Associates of New York, New York, New York